CLINICAL TRIAL: NCT01780246
Title: An Open-label Study to Assess the Safety and Tolerability of a Single Intrathecal Dose of ISIS 396443 in Patients With Spinal Muscular Atrophy Who Previously Participated in ISIS 396443-CS1
Brief Title: An Open-label Safety and Tolerability Study of Nusinersen (ISIS 396443) in Participants With Spinal Muscular Atrophy Who Previously Participated in ISIS 396443-CS1 (NCT01494701)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 396443-CS10
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; SMA; SMN; SMNRx; ISIS-SMNRx; ISIS 396443
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nusinersen (Experimental)
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — Administered by intrathecal (IT) injection
  Other Names: Sprinraza; ISIS 396443; IONIS-SMN Rx; BIIB058

SUMMARY:
The primary objective of this study is to examine the safety and tolerability of nusinersen (ISIS 396443) administered intrathecally to participants with Spinal Muscular Atrophy (SMA) who previously participated in ISIS 396443-CS1 (NCT02865109). The secondary objective was to examine the plasma pharmacokinetics of a single dose of ISIS 396443 administered intrathecally to participants with SMA who previously participated in ISIS 396443-CS1.

DETAILED DESCRIPTION:
This study was conducted and the protocol was registered by Ionis Pharmaceuticals, Inc.

In August 2016, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical signs attributable to Spinal Muscular Atrophy
* Satisfactory completion of dosing and all study visits in ISIS 396443-CS1 (NCT01494701) with an acceptable safety profile, per Investigator judgement.
* Able to complete all study procedures, measurements and visits and parent/participant has adequately supportive psychosocial circumstances, in the opinion of the investigator
* Estimated life expectancy > 2 years from Screening
* Meets age-appropriate institutional criteria for use of anesthesia/sedation, if use is planned for study procedure

Key Exclusion Criteria:

* Have any new or worsening of existing condition which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the participant participating in or completing the study.
* Dosing in ISIS 396443-CS1 (NCT01494701) within 270 days (9 months) of screening, or longer ago than 450 days (15 months)
* Dosing in ISIS 396443-CS2 (NCT01703988)
* Hospitalization for surgery (i.e. scoliosis surgery) or pulmonary event within 2 months of screening or planned during the duration of the study
* Presence of an untreated or inadequately treated active infection requiring systemic antiviral or antimicrobial therapy any time during the screening period
* Clinically significant abnormalities in hematology or clinical chemistry parameters
* Treatment with investigational drug, biological agent, or device within 1-month of Screening or 5 half-lives of study agent, whichever is longer. Treatment with valproate or hydroxyurea within 1 months of screening. Any history of gene therapy or cell transplantation

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience Adverse Events (AEs) and Serious Adverse Events | Up to 24 Weeks
Number of participants with clinically significant neurological examination abnormalities | Up tp 24 Weeks
Number of participants with clinically significant vital sign abnormalities | Up to 24 Weeks
Number of participants with clinically significant physical examination abnormalities | Up to 24 Weeks
Number of participants with clinically significant weight abnormalities | Up to 24 Weeks
Number of participants with clinically significant laboratory parameters | Up to 24 Weeks
Number of participants with clinically significant electrocardiograms (ECGs) abnormalities | Up to 24 Weeks
Number of participants who use concomitant medications | Up to 24 Weeks

SECONDARY OUTCOMES:
PK parameters of nusinersen (ISIS 396443): Maximum observed plasma drug concentration (Cmax) | Plasma at 1, 2, 4 and 6 hours after dosing
PK parameters of nusinersen: Time to reach maximum observed concentration (Tmax) | Plasma at 1, 2, 4 and 6 hours after dosing
PK parameters of nusinersen: Area under the plasma concentrations time curve from the time of the intrathecal (IT) dose to the last collected sample (AUCinf) | Plasma at 1, 2, 4 and 6 hours after dosing
PK parameters of nusinersen (ISIS 396443): Apparent terminal elimination half-life (t1/2), if possible | Plasma at 1, 2, 4 and 6 hours after dosing

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - UT Southwestern Medical Center - Children's Medical Center Dallas, Dallas, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Derived] Darras BT, Farrar MA, Mercuri E, Finkel RS, Foster R, Hughes SG, Bhan I, Farwell W, Gheuens S. An Integrated Safety Analysis of Infants and Children with Symptomatic Spinal Muscular Atrophy (SMA) Treated with Nusinersen in Seven Clinical Trials. CNS Drugs. 2019 Sep;33(9):919-932. doi: 10.1007/s40263-019-00656-w. PMID 31420846
- [Derived] Hache M, Swoboda KJ, Sethna N, Farrow-Gillespie A, Khandji A, Xia S, Bishop KM. Intrathecal Injections in Children With Spinal Muscular Atrophy: Nusinersen Clinical Trial Experience. J Child Neurol. 2016 Jun;31(7):899-906. doi: 10.1177/0883073815627882. Epub 2016 Jan 27. PMID 26823478
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — http://www.rarediseases.org
- See also: Clinical Study Report (CSR) Synopsis - a results summary — http://clinicalresearch.biogen.com/Content/Studies/CS10%20Biogen.com%20Packet.pdf